CLINICAL TRIAL: NCT01363440
Title: A Double-Masked, Randomized, Active-Controlled, Phase 3 Study of the Efficacy and Safety of Intravitreal Administration of VEGF Trap-Eye in Patients With Diabetic Macular Edema
Brief Title: Study of Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) in Patients With Diabetic Macular Edema
Acronym: VISTA DME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VGFT-OD-1009
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Macular Laser Photocoagulation Treatment (Control) (Active Comparator): Participants received macular laser treatment at baseline and as-needed at visits at which laser re-treatment criteria were met, but no more frequently than every 12 weeks.
  Interventions: Procedure: Macular Laser Photocoagulation
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 (Experimental): Participants received 2mg Intravitreal aflibercept injection (IAI) every 4 weeks.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321)
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 (Experimental): Participants received 2mg Intravitreal aflibercept injection (IAI) every 4 weeks for 5 visits followed by injections every 8 weeks.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321)

INTERVENTIONS:
Drug: Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321)
  Arms: Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4; Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Procedure: Macular Laser Photocoagulation — Laser therapy
  Arms: Macular Laser Photocoagulation Treatment (Control)

SUMMARY:
The purpose of this study is to determine the efficacy of Intravitreal Aflibercept Injection (IAI; EYLEA®; BAY86-5321) on the best corrected visual acuity (BCVA) assessed by the early treatment diabetic retinopathy study (ETDRS) chart in patients with diabetic macular edema (DME) with central involvement.

ELIGIBILITY:
Inclusion Criteria:

The following is an abbreviated list of inclusion criteria:

* Adults ≥ 18 years with type 1 or 2 diabetes mellitus
* Decrease in vision determined to be primarily the result of DME in the study eye
* BCVA ETDRS letter score of 73 to 24 (20/40 to 20/320) in the study eye

Exclusion Criteria:

The following is an abbreviated list of exclusion criteria:

* Laser photocoagulation (panretinal or macular) in the study eye within 90 days of day 1
* Previous use of intraocular or periocular corticosteroids in the study eye within 120 days of day 1
* Previous treatment with anti-angiogenic drugs in the study eye (pegaptanib sodium, bevacizumab, ranibizumab, etc.) within 90 days of day 1
* Active proliferative diabetic retinopathy (PDR) in the study eye
* Uncontrolled diabetes mellitus
* Only 1 functional eye even if that eye is otherwise eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (51):
- United States (51):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Arcadia, California
  - Beverly Hills, California
  - La Jolla, California
  - Mountain View, California
  - Oakland, California
  - Palm Desert, California
  - Sacramento, California
  - San Francisco, California
  - Santa Barbara, California
  - Torrance, California
  - Colorado Springs, Colorado
  - Golden, Colorado
  - New London, Connecticut
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Orlando, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - ‘Aiea, Hawaii
  - Wichita, Kansas
  - Portland, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Missoula, Montana
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - Northfield, New Jersey
  - Teaneck, New Jersey
  - Lynbrook, New York
  - Orchard Park, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Portland, Oregon
  - Kingston, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Florence, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Harlingen, Texas
  - Houston, Texas
  - San Antonio (2 Locations), Texas
  - The Woodlands, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Matar K, Indurkar A, Yordi S, Cetin H, Reese JL, Srivastava SK, Ehlers JP. Expanding insights from the VISTA phase III trial: longitudinal comparative assessment of ellipsoid zone integrity and volumetric fluid dynamics. Sci Rep. 2025 Dec 5;15(1):43222. doi: 10.1038/s41598-025-27350-w. PMID 41350590
- [Derived] Dhoot DS, Moini H, Reed K, Silva FQ, Berliner A, Du W, Sharma S. INCIDENCE OF NEW DIABETIC MACULAR EDEMA IN FELLOW EYES OF PATIENTS IN THE VISTA AND VIVID STUDIES. Retina. 2023 Feb 1;43(2):254-262. doi: 10.1097/IAE.0000000000003658. Epub 2022 Oct 17. PMID 36265076
- [Derived] Dhoot DS, Moini H, Reed K, Du W, Vitti R, Berliner AJ, Singh RP. Functional outcomes of sustained improvement on Diabetic Retinopathy Severity Scale with intravitreal aflibercept in the VISTA and VIVID trials. Eye (Lond). 2023 Jul;37(10):2020-2025. doi: 10.1038/s41433-022-02058-7. Epub 2022 Apr 19. PMID 35440699
- [Derived] Wykoff CC, Shah C, Dhoot D, Coleman HR, Thompson D, Du W, Baker K, Vitti R, Berliner AJ, Metzig C, Saroj N. Longitudinal Retinal Perfusion Status in Eyes with Diabetic Macular Edema Receiving Intravitreal Aflibercept or Laser in VISTA Study. Ophthalmology. 2019 Aug;126(8):1171-1180. doi: 10.1016/j.ophtha.2019.03.040. Epub 2019 Apr 1. PMID 30946887
- [Derived] Midena E, Gillies M, Katz TA, Metzig C, Lu C, Ogura Y. Impact of Baseline Central Retinal Thickness on Outcomes in the VIVID-DME and VISTA-DME Studies. J Ophthalmol. 2018 Mar 29;2018:3640135. doi: 10.1155/2018/3640135. eCollection 2018. PMID 29785301
- [Derived] Staurenghi G, Feltgen N, Arnold JJ, Katz TA, Metzig C, Lu C, Holz FG; VIVID-DME and VISTA-DME study investigators. Impact of baseline Diabetic Retinopathy Severity Scale scores on visual outcomes in the VIVID-DME and VISTA-DME studies. Br J Ophthalmol. 2018 Jul;102(7):954-958. doi: 10.1136/bjophthalmol-2017-310664. Epub 2017 Oct 19. PMID 29051325
- [Derived] Wykoff CC, Marcus DM, Midena E, Korobelnik JF, Saroj N, Gibson A, Vitti R, Berliner AJ, Williams Liu Z, Zeitz O, Metzig C, Schmelter T, Heier JS. Intravitreal Aflibercept Injection in Eyes With Substantial Vision Loss After Laser Photocoagulation for Diabetic Macular Edema: Subanalysis of the VISTA and VIVID Randomized Clinical Trials. JAMA Ophthalmol. 2017 Feb 1;135(2):107-114. doi: 10.1001/jamaophthalmol.2016.4912. PMID 28006063
- [Derived] Ziemssen F, Schlottman PG, Lim JI, Agostini H, Lang GE, Bandello F. Initiation of intravitreal aflibercept injection treatment in patients with diabetic macular edema: a review of VIVID-DME and VISTA-DME data. Int J Retina Vitreous. 2016 Jul 11;2:16. doi: 10.1186/s40942-016-0041-z. eCollection 2016. PMID 27847634

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with diabetic macular edema (DME) secondary to diabetes mellitus involving the center of the macula in the study eye could participate in the study.
Pre-assignment Details: Of 687 participants who were screened for inclusion in the study, 466 were enrolled (started) and 461 received treatment.
Period: Overall Study
Arm/Group | Macular Laser Photocoagulation Treatment (Control) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Started | 156 (randomized) | 156 (randomized) | 154 (randomized)
Participants Received Treatment | 154 (safety analysis set (SAF)) | 155 (safety analysis set (SAF)) | 152 (safety analysis set (SAF))
Completed Week 52 | 145 | 146 | 144
Completed Week 100 | 133 | 125 | 127
Completed | 133 (Completed Week 100) | 125 (Completed Week 100) | 127 (Completed Week 100)
Not Completed | 23 | 31 | 27
Not completed — Adverse Event | 5 | 4 | 4
Not completed — Death | 3 | 7 | 5
Not completed — Withdrawal by Subject | 9 | 11 | 11
Not completed — Lost to Follow-up | 2 | 4 | 5
Not completed — Other | 4 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Baseline population analyzed using the SAF
Groups:
- Control: Participants received macular laser treatment at baseline and as-needed at visits at which laser re-treatment criteria were met, but no more frequently than every 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Control | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Total
Number analyzed (Participants) | 154 | 155 | 152 | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.65) | 62 (11.16) | 63.1 (9.36) | 62.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 73 | 210
  Male | 85 | 87 | 79 | 251

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 52 - Last Observation Carried Forward (LOCF)
Description: Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of 73 to 24 (= Acuity of 20/40 to 20/320) in the study eye were included; a higher score represents better functioning.
Time Frame: Baseline and Week 52
Population: The Primary efficacy endpoint was analyzed using the full analysis set (FAS). The FAS included all 'Participants received Treatment' and had a baseline and at least 1 post-baseline assessment of Best Corrected Visual Acuity (BCVA).
Measure: Least Squares Mean (Standard Error); unit: letters correctly read
Arm/Group | Control | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Number analyzed (Participants) | 154 | 154 | 151
letters correctly read | .10 (1.03) | 12.3 (.76) | 10.6 (.69)
Statistical Analysis 1: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Net) = 12.19, 97.5% CI 2-sided [9.35 to 15.04]
Statistical Analysis 2: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Net) = 10.45, 97.5% CI 2-sided [7.73 to 13.17]

2. Secondary Outcome: Percentage of Participants Who Gained at Least 10 Letters in BCVA as Measured by ETDRS Letter Score Compared With Baseline at Week 52 - LOCF
Time Frame: Baseline and Week 52
Population: All secondary efficacy endpoints were analyzed using the full analysis set (FAS). The FAS included all 'Participants received Treatment' and had a baseline and at least 1 post-baseline assessment of Best Corrected Visual Acuity (BCVA).
Measure: Number; unit: percentage of participants
Arm/Group | Control | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Number analyzed (Participants) | 154 | 154 | 151
percentage of participants | 30 | 100 | 88
Statistical Analysis 1: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4; Test type: Superiority or Other; p = .0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 45.9, 97.5% CI 2-sided [34.7 to 57.0]
Statistical Analysis 2: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8; Test type: Superiority or Other; p = .0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 38.8, 97.5% CI 2-sided [27.2 to 50.3]

3. Secondary Outcome: Percentage of Participants Who Gained at Least 15 Letters in BCVA as Measured by ETDRS Letter Score Compared With Baseline at Week 52 - LOCF
Time Frame: Baseline and Week 52
Measure: Number; unit: percentage of participants
Arm/Group | Control | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Number analyzed (Participants) | 154 | 154 | 151
percentage of participants | 12 | 64 | 47
Statistical Analysis 1: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 34.2, 97.5% CI 2-sided [24.1 to 44.4]
Statistical Analysis 2: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 23.3, 97.5% CI 2-sided [13.5 to 33.1]

4. Secondary Outcome: Percentage of Participants With a ≥2-step Improvement From Baseline in the ETDRS DRSS (Diabetic Retinopathy Severity Score) as Assessed by FP (Fundus Photography) at Week 52 - LOCF
Description: Baseline ETDRS DRSS: None (level 10); Mild to moderate nonproliferative DR (levels 14, 15, 20, 35, and 43); Moderately severe/severe nonproliferative DR (levels 47 and 53); Mild/moderate/high-risk/advanced proliferative DR (levels 61, 65, 71,75, 81, and 85)
Time Frame: Baseline and Week 52
Measure: Number; unit: percentage of participants
Arm/Group | Control | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Number analyzed (Participants) | 154 | 154 | 151
percentage of participants | 22 | 52 | 44
Statistical Analysis 1: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 19.7, 97.5% CI 2-sided [9.0 to 30.4]
Statistical Analysis 2: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8; Test type: Superiority or Other; p = 0.0017, Cochran-Mantel-Haenszel; Mean Difference (Net) = 14.9, 97.5% CI 2-sided [4.4 to 25.4]

5. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) at Week 52 as Assessed on Optical Coherence Tomography (OCT) - LOCF
Time Frame: Baseline and Week 52
Measure: Least Squares Mean (Standard Error); unit: microns
Arm/Group | Control | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Number analyzed (Participants) | 154 | 154 | 151
microns | -73.3 (12.09) | -184.1 (6.57) | -186.8 (6.90)
Statistical Analysis 1: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Net) = -110.8, 97.5% CI 2-sided [-141.3 to -80.22]
Statistical Analysis 2: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Net) = -113.5, 97.5% CI 2-sided [-144.2 to -82.75]

6. Secondary Outcome: Change From Baseline in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Near Activities Subscale at Week 52 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales that are all scored from 0-100. Near activities are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf.
Time Frame: Baseline and Week 52
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Control | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Number analyzed (Participants) | 154 | 154 | 151
scores on a scale | 3.7 (1.55) | 8.9 (1.58) | 8.1 (1.44)
Statistical Analysis 1: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4; Test type: Superiority or Other; p = 0.0168, ANCOVA; Mean Difference (Net) = 5.19, 97.5% CI [0.33 to 10.04]
Statistical Analysis 2: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8; Test type: Superiority or Other; p = 0.0323, ANCOVA; Mean Difference (Net) = 4.36, 97.5% CI 2-sided [-0.21 to 8.93]

7. Secondary Outcome: Change From Baseline in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Distance Activities Subscale at Week 52 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales that are all scored from 0-100. Distance activities are defined as reading street signs or names on stores, and going down stairs, steps, or curbs.
Time Frame: Baseline and Week 52
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Control | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8
Number analyzed (Participants) | 154 | 154 | 151
scores on a scale | 4.9 (1.44) | 7.7 (1.57) | 6.5 (1.48)
Statistical Analysis 1: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4; Test type: Superiority or Other; p = 0.1702, ANCOVA; Mean Difference (Net) = 2.86, 97.5% CI 2-sided [-1.82 to 7.54]
Statistical Analysis 2: Comparison: Control vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8; Test type: Superiority or Other; p = 0.4067, ANCOVA; Mean Difference (Net) = 1.65, 97.5% CI 2-sided [-2.83 to 6.13]

ADVERSE EVENTS:
Time Frame: From the first study drug injection until 30 days after the last study drug injection at the latest from week 0 to week 100; From the first study drug injection until 30 days after the last study drug injection at the latest from week 0 to week 148.
Groups:
- Control (Week 0 to Week 100); Control (Week 0 to Week 148): Participants received macular laser treatment at baseline and as-needed at visits at which laser re-treatment criteria were met, but no more frequently than every 12 weeks.
- IAI;EYLEA®;BAY86-5321 2Q4 (Week 0 to Week 100): Participants received 2mg Intravitreal aflibercept injection (IAI) every 4 weeks.
- IAI;EYLEA®;BAY86-5321) 2Q8 (Week 0 to Week 100); IAI;EYLEA®;BAY86-5321) 2Q8 (Week 0 to Week 148): Participants received 2mg Intravitreal aflibercept injection (IAI) every 4 weeks for 5 visits followed by injections every 8 weeks.
- IAI;EYLEA®;BAY86-5321 2Q4 (Week 0 to Week 148): Participants received 2mg Intravitreal aflibercept injection(IAI) every 4 weeks.
Arm/Group | Control (Week 0 to Week 100) | IAI;EYLEA®;BAY86-5321 2Q4 (Week 0 to Week 100) | IAI;EYLEA®;BAY86-5321) 2Q8 (Week 0 to Week 100) | Control (Week 0 to Week 148) | IAI;EYLEA®;BAY86-5321 2Q4 (Week 0 to Week 148) | IAI;EYLEA®;BAY86-5321) 2Q8 (Week 0 to Week 148)
Serious Adverse Events (participants affected / at risk) | 67/154 | 67/155 | 56/152 | 84/154 | 85/155 | 75/152
Other Adverse Events (participants affected / at risk) | 91/154 | 90/155 | 76/152 | 134/154 | 137/155 | 136/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (Week 0 to Week 100) (N=154) | IAI;EYLEA®;BAY86-5321 2Q4 (Week 0 to Week 100) (N=155) | IAI;EYLEA®;BAY86-5321) 2Q8 (Week 0 to Week 100) (N=152) | Control (Week 0 to Week 148) (N=154) | IAI;EYLEA®;BAY86-5321 2Q4 (Week 0 to Week 148) (N=155) | IAI;EYLEA®;BAY86-5321) 2Q8 (Week 0 to Week 148) (N=152)
Anaemia (Blood and lymphatic system disorders) | 1 | 9 | 5 | 2 | 10 | 6
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 2 | 2 | 4 | 2 | 3
Angina pectoris (Cardiac disorders) | 1 | 1 | 1 | 1 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 3 | 0 | 2 | 4
Atrial flutter (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 1 | 3 | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 4 | 1 | 0 | 4 | 2 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 5 | 9 | 5 | 6 | 11 | 6
Cor pulmonale chronic (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 4 | 2 | 2 | 5 | 4
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 3 | 4 | 5 | 3 | 4 | 5
Coronary ostial stenosis (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 5 | 3 | 3 | 4 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Systolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 1
Cataract (Eye disorders) | 1 | 4 | 0 | 1 | 4 | 0 — Study eye
Cataract subcapsular (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cataract subcapsular (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Study eye
Corneal epithelium defect (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 — Study eye
Diabetic retinal oedema (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Diabetic retinal oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Study eye
Diabetic retinopathy (Eye disorders) | 2 | 0 | 0 | 2 | 0 | 0 — Study eye
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyphaema (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Study eye
Intraocular pressure increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Iris neovascularisation (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Lens dislocation (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Study eye
Macular ischaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Study eye
Punctate keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Study eye
Retinal aneurysm (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Study eye
Retinal detachment (Eye disorders) | 1 | 2 | 1 | 2 | 3 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 0 — Study eye
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Study eye
Retinal haemorrhage (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 0
Retinal ischaemia (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 — Study eye
Retinal ischaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 — Study eye
Retinal neovascularisation (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 1
Retinal vascular disorder (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 — Study eye
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 1 | 0 | 1 | 1 — Study eye
Vitreous haemorrhage (Eye disorders) | 3 | 2 | 1 | 3 | 3 | 2 — Study eye
Vitreous haemorrhage (Eye disorders) | 2 | 7 | 2 | 3 | 9 | 4
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 3 | 9 | 4
Vitreous opacities (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3 | 1 | 2 | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Internal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0 | 2
Chest pain (General disorders) | 3 | 1 | 4 | 4 | 1 | 4
Death (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Device failure (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Device malfunction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Medical device complication (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 1 | 2 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 2 | 0 | 1
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 2 | 2 | 2 | 2 | 2 | 2
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 1 | 2 | 1
Burn infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 4 | 7 | 8 | 5 | 9 | 8
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 — Study eye
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 2 | 1 | 2 | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 1 | 2 | 1 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1 | 0 | 1 | 3 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 3 | 5 | 2 | 5 | 7 | 3
Osteomyelitis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 4 | 3 | 4 | 6 | 4
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 2 | 0 | 2 | 3 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 4 | 2 | 1
Urosepsis (Infections and infestations) | 1 | 2 | 1 | 1 | 2 | 1
Wound sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Clavical fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 5 | 3 | 3 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1 | 2 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 — Study eye
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity tests abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 — Study eye
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2 | 4 | 2 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0 | 4 | 2
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 2 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 3 | 1 | 6 | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 5 | 0 | 1 | 6 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Ketosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 3 | 5 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Tendonitits (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 3 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Diffuse large B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 0 | 1 | 3
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 3 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0 | 1 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Brain stem stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 2 | 0 | 0 | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 5 | 5 | 4 | 5 | 5
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 2 | 1 | 1
Diabetic coma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sedation (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 2 | 0 | 3 | 3 | 1
Thalamic infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 0 | 1 | 3 | 1 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Study eye
Affective disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 1 | 0 | 2 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2 | 1 | 0 | 2 | 1
Schizoaffective disorder (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Intercapillary glomerulosclerosis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrosclerosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 4 | 5 | 1 | 5 | 5 | 1
Renal failure acute (Renal and urinary disorders) | 7 | 6 | 6 | 9 | 10 | 8
Renal failure chronic (Renal and urinary disorders) | 2 | 4 | 3 | 4 | 5 | 3
Renal impairment (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Labia enlarged (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1
Uterine mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 3 | 2
Hypertrophic scar (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Foot amputation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 5 | 1 | 3 | 6 | 2
Hypertensive crisis (Vascular disorders) | 2 | 2 | 0 | 2 | 2 | 0
Hypertensive emergency (Vascular disorders) | 1 | 1 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 1 | 0 | 2 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (Week 0 to Week 100) (N=154) | IAI;EYLEA®;BAY86-5321 2Q4 (Week 0 to Week 100) (N=155) | IAI;EYLEA®;BAY86-5321) 2Q8 (Week 0 to Week 100) (N=152) | Control (Week 0 to Week 148) (N=154) | IAI;EYLEA®;BAY86-5321 2Q4 (Week 0 to Week 148) (N=155) | IAI;EYLEA®;BAY86-5321) 2Q8 (Week 0 to Week 148) (N=152)
Anaemia (Blood and lymphatic system disorders) | 12 | 20 | 12 | 15 | 27 | 20
Anxiety (Psychiatric disorders) | 7 | 12 | 4 | 9 | 13 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 8 | 8 | 12 | 13 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 5 | 10 | 7 | 6 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 20 | 6 | 11 | 22 | 9
Blood creatine phosphokinase increased (Investigations) | 12 | 7 | 4 | 12 | 9 | 4
Blood glucose increased (Investigations) | 6 | 9 | 11 | 9 | 15 | 16
Blood pressure increased (Investigations) | 10 | 9 | 7 | 15 | 12 | 8
Blood pressure systolic increased (Investigations) | 2 | 2 | 5 | 2 | 4 | 8
Bronchitis (Infections and infestations) | 11 | 12 | 4 | 13 | 12 | 7
Cardiac failure congestive (Cardiac disorders) | 6 | 12 | 9 | 4 | 6 | 8
Cataract (Eye disorders) | 17 | 15 | 11 | 25 | 22 | 17
Cataract (Eye disorders) | 16 | 21 | 13 | 24 | 28 | 21 — Study eye
Cataract cortical (Eye disorders) | 6 | 3 | 6 | 11 | 2 | 7 — Study eye
Cataract cortical (Eye disorders) | 8 | 2 | 7 | 8 | 5 | 7
Cataract nuclear (Eye disorders) | 2 | 6 | 2 | 6 | 8 | 3 — Study eye
Cataract nuclear (Eye disorders) | 2 | 6 | 2 | 2 | 8 | 2
Cataract subcapsular (Eye disorders) | 6 | 4 | 8 | 8 | 8 | 10
Cataract subcapsular (Eye disorders) | 7 | 6 | 8 | 10 | 12 | 10 — Study eye
Cellulitis (Infections and infestations) | 7 | 10 | 12 | 7 | 5 | 8
Chest pain (General disorders) | 9 | 3 | 5 | 9 | 3 | 5
Conjunctival haemorrhage (Eye disorders) | 29 | 30 | 27 | 31 | 35 | 29
Conjunctival haemorrhage (Eye disorders) | 53 | 63 | 48 | 55 | 63 | 50 — Study eye
Constipation (Gastrointestinal disorders) | 9 | 11 | 5 | 14 | 15 | 6
Corneal abrasion (Eye disorders) | 6 | 4 | 6 | 9 | 7 | 6 — Study eye
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 18 | 17 | 16 | 21 | 20
Depression (Psychiatric disorders) | 7 | 7 | 4 | 9 | 6 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 20 | 13 | 19 | 28 | 23 | 25
Diabetic retinal oedema (Eye disorders) | 19 | 22 | 18 | 26 | 29 | 23
Diabetic retinopathy (Eye disorders) | 11 | 8 | 14 | 16 | 8 | 18
Diarrhoea (Gastrointestinal disorders) | 13 | 14 | 6 | 15 | 19 | 7
Dizziness (Nervous system disorders) | 8 | 7 | 9 | 9 | 9 | 10
Drug hypersensitivity (Immune system disorders) | 2 | 5 | 3 | 6 | 8 | 3
Dry eye (Eye disorders) | 7 | 12 | 7 | 8 | 13 | 9
Dry eye (Eye disorders) | 10 | 14 | 7 | 12 | 16 | 9 — Study eye
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 12 | 11 | 7 | 15 | 13
Ear infection (Infections and infestations) | 4 | 3 | 6 | 6 | 5 | 9
Eye irritation (Eye disorders) | 12 | 15 | 11 | 14 | 15 | 13 — Study eye
Eye irritation (Eye disorders) | 7 | 6 | 7 | 8 | 9 | 8
Eye pain (Eye disorders) | 20 | 23 | 21 | 23 | 23 | 26 — Study eye
Eye pain (Eye disorders) | 7 | 11 | 9 | 10 | 13 | 14
Fall (Injury, poisoning and procedural complications) | 8 | 7 | 12 | 12 | 7 | 14
Fatigue (General disorders) | 4 | 8 | 3 | 5 | 9 | 3
Foreign body sensation in eyes (Eye disorders) | 8 | 8 | 5 | 8 | 9 | 6 — Study eye
Gastroenteritis viral (Infections and infestations) | 2 | 2 | 6 | 2 | 3 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 10 | 4 | 14 | 13 | 10
Glycosylated haemoglobin increased (Investigations) | 7 | 7 | 13 | 10 | 10 | 16
Headache (Nervous system disorders) | 19 | 18 | 7 | 22 | 21 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 5 | 3 | 13 | 6 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 9 | 6 | 9 | 11 | 8
Hypertension (Vascular disorders) | 49 | 41 | 42 | 56 | 51 | 49
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 8 | 5 | 10 | 14 | 9
Hypothyroidism (Endocrine disorders) | 7 | 4 | 5 | 8 | 4 | 5
Influenza (Infections and infestations) | 9 | 7 | 16 | 15 | 9 | 22
Intraocular pressure increased (Investigations) | 2 | 12 | 10 | 6 | 16 | 10 — Study eye
Lacrimation increased (Eye disorders) | 3 | 4 | 7 | 4 | 5 | 9
Lacrimation increased (Eye disorders) | 6 | 7 | 6 | 7 | 8 | 8 — Study eye
Localised infection (Infections and infestations) | 5 | 10 | 5 | 11 | 11 | 5
Macular fibrosis (Eye disorders) | 15 | 11 | 15 | 20 | 13 | 17 — Study eye
Macular fibrosis (Eye disorders) | 12 | 11 | 16 | 19 | 14 | 23
Macular oedema (Eye disorders) | 1 | 4 | 6 | 7 | 6 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 5 | 2 | 9 | 6 | 4
Nasopharyngitis (Infections and infestations) | 17 | 17 | 19 | 23 | 22 | 24
Nausea (Gastrointestinal disorders) | 15 | 19 | 11 | 16 | 21 | 16
Neuropathy peripheral (Nervous system disorders) | 5 | 5 | 7 | 6 | 6 | 8
Ocular hyperaemia (Eye disorders) | 12 | 6 | 6 | 12 | 6 | 7 — Study eye
Oedema peripheral (General disorders) | 8 | 15 | 15 | 11 | 19 | 16
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 7 | 5 | 6 | 4 | 12
Pain in extremity (Eye disorders) | 10 | 8 | 5 | 13 | 12 | 7
Photopsia (Eye disorders) | 7 | 2 | 1 | 8 | 2 | 2 — Study eye
Pneumonia (Infections and infestations) | 7 | 8 | 7 | 4 | 9 | 6
Posterior capsule opacification (Eye disorders) | 10 | 5 | 5 | 12 | 8 | 10
Posterior capsule opacification (Eye disorders) | 12 | 7 | 8 | 16 | 9 | 15 — Study eye
Procedural pain (Injury, poisoning and procedural complications) | 1 | 8 | 2 | 2 | 8 | 3
Punctate keratitis (Eye disorders) | 1 | 5 | 7 | 3 | 8 | 7 — Study eye
Pyrexia (General disorders) | 2 | 7 | 6 | 5 | 10 | 7
Renal failure acute (Renal and urinary disorders) | 11 | 10 | 9 | 5 | 8 | 7
Renal failure chronic (Renal and urinary disorders) | 4 | 9 | 8 | 5 | 9 | 8
Retinal exudates (Eye disorders) | 13 | 12 | 4 | 14 | 15 | 6 — Study eye
Retinal exudates (Eye disorders) | 11 | 12 | 6 | 15 | 15 | 8
Retinal haemorrhage (Eye disorders) | 15 | 10 | 5 | 16 | 13 | 7 — Study eye
Retinal haemorrhage (Eye disorders) | 10 | 11 | 5 | 13 | 16 | 6
Retinal neovascularisation (Eye disorders) | 10 | 10 | 4 | 12 | 10 | 5
Retinal neovascularisation (Eye disorders) | 12 | 3 | 3 | 12 | 3 | 3 — Study eye
Retinal pigment epitheliopathy (Eye disorders) | 3 | 5 | 8 | 3 | 6 | 9 — Study eye
Seasonal allergy (Immune system disorders) | 8 | 6 | 9 | 9 | 9 | 12
Sinusitis (Infections and infestations) | 12 | 13 | 12 | 18 | 14 | 13
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 6 | 9 | 5 | 9 | 12 | 6
Upper respiratory tract infection (Infections and infestations) | 13 | 11 | 15 | 16 | 13 | 17
Urinary tract infection (Infections and infestations) | 14 | 17 | 26 | 20 | 30 | 32
Urine protein/ creatinine ratio increased (Investigations) | 8 | 5 | 2 | 9 | 8 | 3
Vision blurred (Eye disorders) | 10 | 11 | 6 | 13 | 14 | 9 — Study eye
Vision blurred (Eye disorders) | 5 | 8 | 5 | 7 | 11 | 7
Visual Impairment (Eye disorders) | 7 | 1 | 3 | 8 | 1 | 3 — Study eye
Visual acuity reduced (Eye disorders) | 6 | 4 | 10 | 10 | 8 | 10
Visual acuity reduced (Eye disorders) | 11 | 7 | 10 | 14 | 10 | 12 — Study eye
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 | 6 | 5 | 7 | 8 | 7
Vitreous detachment (Eye disorders) | 16 | 15 | 18 | 23 | 17 | 23
Vitreous detachment (Eye disorders) | 15 | 14 | 22 | 20 | 20 | 25 — Study eye
Vitreous floaters (Eye disorders) | 10 | 11 | 10 | 12 | 15 | 14
Vitreous floaters (Eye disorders) | 14 | 21 | 17 | 16 | 23 | 21 — Study eye
Vitreous haemorrhage (Eye disorders) | 12 | 9 | 2 | 13 | 10 | 4 — Study eye
Vitreous haemorrhage (Eye disorders) | 11 | 8 | 5 | 19 | 11 | 7
Vomiting (Gastrointestinal disorders) | 7 | 14 | 3 | 9 | 16 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission of any (M)anuscript, (I)nstitution shall, or cause PI to, provide (S)ponsor a copy of (M). (I) to consider comments submitted by (S), & to delete confidential information upon (S) request. At (S)'s request, (I) to delay publication for an additional 60 days to allow filing of patent applications. (I) & PI agree to delay publication, prior to (M) summarizing data from all sites, unless no (M) is published prior to first anniversary of final study report.